CLINICAL TRIAL: NCT01546090
Title: Effect of Preoperative Alprazolam on the Success of Inferior Alveolar Nerve Block for Teeth With Irreversible Pulpitis
Brief Title: Effect of Alprazolam on the Success of Inferior Alveolar Nerve (IAN) Block
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Isfahan University of Medical Sciences (Other)
Collaborators: University of Isfahan (Other)
Responsible Party: Principal Investigator, Masoud Saatchi, Associate Professor of Endodontics, Isfahan University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 390553; 390553; 390553 (Other: School of Dentistry)
Record Dates: First submitted 2012-03-02; First posted 2012-03-07 (Estimated); Last update posted 2012-03-07 (Estimated); Status verified 2012-03

CONDITIONS: Inferior Alveolar Nerve Block Failure
Keywords: Alprazolam; benzodiazepines; Inferior alveolar nerve block; irreversible pulpitis; local anesthesia
MeSH Terms: interventions — Alprazolam; Starch

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- alprazolam (Experimental): Alprazolam is a short-acting anxiolytic of the benzodiazepine class of psychoactive drugs
  Interventions: Drug: Alprazolam
- placebo (Placebo Comparator): placebo capsules were filled with starch
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Alprazolam — preoperative administration of an orally 0.50 mg single dose
  Other Names: xanax, Pfizer
  Arms: alprazolam
Drug: placebo — placebo capsules were filled with starch
  Other Names: starch
  Arms: placebo

SUMMARY:
The purpose of this prospective, randomized, double-blind, placebo-controlled study is to evaluate the effect of preoperative administration of alprazolam on the success of the IAN block for teeth with irreversible pulpitis.

DETAILED DESCRIPTION:
Sixty patients diagnosed with irreversible pulpitis of a mandibular molar randomly receive, in a double-blind manner, identical capsules of either 0.50 mg alprazolam or placebo 45 minutes before the administration of a conventional IAN block. Access is begun 15 minutes after completion of the IAN block, and all patients profound lip numbness. Success is defined as no or mild pain based on visual analog scale recordings during access preparation and initial instrumentation.

ELIGIBILITY:
Inclusion Criteria:

* patients with active pain in a mandibular molar
* prolonged response to cold testing with Endo-Frost cold spray
* Absence of any periapical radiolucency on radiographs
* a vital pulp while access cavity preparation
* ability to understand the use of pain scales.

Exclusion Criteria:

* patients were having allergy and sensitivity to benzodiazepines
* pregnant and breast feeding patients
* patients who had taken sedation within 24 hours before the treatment
* having pain in more than one mandibular tooth
* unable to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-03; Primary Completion 2011-10 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
the success rate of the IAN block | one hour after administration of alprazolam

SECONDARY OUTCOMES:
initial pain | one hour after administration of alprazolam

CONTACTS AND LOCATIONS:
Locations (1):
- School of Dentistry, Isfahan University of Medical Sciences, Isfahan, Isfahan, Iran

REFERENCES:
- [Result] Lindemann M, Reader A, Nusstein J, Drum M, Beck M. Effect of sublingual triazolam on the success of inferior alveolar nerve block in patients with irreversible pulpitis. J Endod. 2008 Oct;34(10):1167-70. doi: 10.1016/j.joen.2008.07.013. Epub 2008 Aug 23. PMID 18793913